CLINICAL TRIAL: NCT05452629
Title: Effect of Brief Mindfulness and Relaxation Inductions on Anxiety, Affect and Brain Activation in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PACNL_JT_MI_EEG
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: State Anxiety; Affect; Electroencephalography
Keywords: Mindfulness; Relaxation; Mental health; EEG; Cognitive resource
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: In a counterbalanced order, participants completed three conditions that incorporated two 30-minute experimental conditions (i.e., MI or RI) and a control condition (i.e., opened thinking)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness Induction (Experimental): A brief and single session of mindfulness practice for 30-minute.
  Interventions: Behavioral: Mindfulness induction (MI)
- Relaxation Induction (Experimental): A brief and single session of self-directed relaxation for 30-minute.
  Interventions: Behavioral: Relaxation (RI)
- Control Condition (No Intervention): Open thinking.

INTERVENTIONS:
Behavioral: Mindfulness induction (MI) — In the MI condition, participants were guided to focus on present experiences regarding the thoughts, emotions and sensations through the three classic mindfulness exercises (i.e., focused breathing, meditation, and body scanning). The duration of MI was 30-minutes.
  Arms: Mindfulness Induction
Behavioral: Relaxation (RI) — In the RI condition, participants were guided to relax each muscle group following the audio for 30-minutes.
  Arms: Relaxation Induction

SUMMARY:
The athlete population has a high risk of suffering from mental health problems (e.g., anxiety), especially for athletes with individual sports. As such, various forms of mental training were used to maintain the mental health of athletes, such as mindfulness training or relaxation training. However, differences pertaining to the electrophysiological mechanisms resulting from both mental training in athletes are unknown. Therefore, the purpose of the current study was to examine the differential effects between the brief mindfulness induction (MI) and relaxation induction (RI) on state anxiety, affect and the activation of the brain in track and field athletes.

DETAILED DESCRIPTION:
The purposes of this study are: (1) examining the effect of brief mindfulness induction (MI) and relaxation induction (RI) on anxiety and affect in athletes with individual sports, (2) and we sought to identify the different brain activity (i.e., theta, alpha) changes between MI and RI using EEG. In the present study, subjects were contrasted using a within-subject comparison across MI, RI, and control condition. According to past works on the comparison of mindfulness and psychological skill training, we hypothesized that MI and RI would both improve anxiety and affect, compared with control condition. Furthermore, we also hypothesized that RI would elicit greater theta power (i.e., more cognitive control) than MI. In addition, when compared with control condition, participants might be elicited greater alpha power during the MI and RI.

ELIGIBILITY:
Inclusion Criteria:

1. track and field athletes with regular training
2. right-handedness
3. no history of neurological illness
4. no regular training experience in mindfulness or relaxation interventions

Exclusion Criteria:

-

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
State anxiety | 10 minutes
  The Chinese version of the State-Trait Anxiety Inventory (C-STAI, Wang & Chung, 2016), which is based on the State-Trait Anxiety Inventory (STAI, Spielberger, 1970), was utilized to assess an individual's alteration of state anxiety before and after each experimental manipulation in current study. The State Anxiety Inventory (SAI) is a 20-item sub-scales in the STAI, with a 4-point Likert scale ranging from 1 (not at all) to 4 (very much so) used for each item. Higher total scores indicate higher levels of state anxiety.
Affective state | 5 minutes
  The Positive and Negative Affect Schedule (PANAS) was utilized to assess an individual's alteration of PA and NA before and after each experimental manipulation in current study. PANAS is a 20-items questionnaire that consists of two 10-item mood scales assessing the positively affective states (i.e., PA) and negatively affective states (i.e., NA), respectively. Participants were asked to rate to what extent they felt a certain way right now from 1 (not at all) to 5 (extremely). Higher total scores indicate higher intensity of affective state.
EEG | 30 minutes
  The selected frequency bands were as theta (4-8 Hz) and alpha (8-13 Hz), the frequency bands were computed by averaged across epochs and integrated spectral power, the frontal region (Fp1, Fp2, F7, F3, Fz, F4, F8) for theta power, and posterior region (P7, P3, Pz, P4, P8, O1, Oz, O2) for alpha power were selected into the statistical analysis, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kai Chang, Ph.D., Study Director — Department of Physical Education and Sport Sciences, National Taiwan Normal University
Locations (1):
- Yu-Kai Chang, Ph.D., Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No